CLINICAL TRIAL: NCT05976022
Title: Personalized Brain Functional Sector-guided rTMS Therapy Over Different Targets for Treatment-resistant Depression
Brief Title: pBFS Guided rTMS Therapy Over Different Targets for Treatment-Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changping Laboratory (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPLMDDdiffTarg_HN
Record Dates: First submitted 2023-07-14; First posted 2023-08-04 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-08

CONDITIONS: MDD; Major Depressive Disorder; Treatment Resistant Depression
Keywords: MDD; Major Depressive Disorder; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- active rTMS (Experimental): 2 sessions with 1800 pulses per session and 50min inter-session interval of active rTMS will deliver to the assigned target
  Interventions: Device: active rTMS

INTERVENTIONS:
Device: active rTMS — 2 sessions with 1800 pulses per session and 50min inter-session interval of active rTMS will deliver to the assigned target

SUMMARY:
To explore the effectiveness and safety of rTMS intervention with different targets in the left prefrontal cortex defined using the pBFS method, in adult patients with moderate and severe depressive disorder. Second, investigate the neural circuit that responds to the rTMS intervention using individualized brain image analysis, which may help to establish an effective target for the neuromodulation of patients with major depressive disorder.

DETAILED DESCRIPTION:
Stimulation of the dorsolateral prefrontal cortex(DLPFC) and ventromedial prefrontal cortex (DMPFC) as target sites for rTMS intervention in depressive disorders has shown some therapeutic efficacy. However, overall patient response rates remain suboptimal, partly because the prefrontal cortex is a large region encompassing multiple functional networks. Analyses suggest that targeting different targets within the dorsolateral and ventromedial prefrontal cortex for intervention in depressive disorder patients may activate distinct functional networks. Therefore, selecting appropriate targets within the prefrontal cortex that accurately modulate the functional networks involved in depressive disorder patients is crucial for achieving effective clinical outcomes. Fox et al. have demonstrated that clinical response and individualized target sites in the dorsolateral prefrontal cortex are associated with functional connectivity to the subgenual cingulate cortex (sgACC). However, some analyses have indicated that rTMS target sites based solely on minimal sgACC connectivity may not be optimal for all depressive symptoms. Therefore, identifying individualized stimulation targets that improve core symptoms in depressed patients is important for achieving more effective personalized treatment of depressive disorders. This study aims to explore the efficacy and safety of rTMS interventions targeting 40 prefrontal cortex sites in depressive disorder patients and functional imaging-based mechanisms for optimal stimulation targets.

After being informed about the study and potential risks. All patients giving written informed consent will undergo a screening period to determine eligibility for study entry. At week 0, patients who meet the eligibility requirements will be assigned a random intervention target from 40 prefrontal cortex sites. Then all participants will undergo a 14-day rTMS modulation and a week follow-up visit. Participants will keep a stable treatment regime during treatment and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of DSM-5(Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) for depression disorder without psychotic symptoms, and currently experiencing a recurrence episode.
* Total HAMD17 score ≥20 and total MADRS score ≥20 before randomization.
* Hospitalized/outpatient patients aged 18-65 years (inclusive), male or female.
* Inadequate response to at least one antidepressant trial of adequate doses and duration.
* A stable antidepressant regimen for at least 4 weeks at a dose not lower than the prescribed range of drug use before randomization.
* The Maudsley Staging Method (MSM) is used to assess patients as having at least a moderate level of treatment-resistant condition (MSM score ≥ 7 points).
* Voluntarily participate in the trial and sign informed consent. Able to comply with the planned visit, examination and treatment plan, and other study procedures.

Exclusion Criteria:

* Meet DSM-5 diagnostic criteria for other mental disorders (such as schizophrenia spectrum disorders, bipolar and related disorders, neurodevelopmental disorders, neurocognitive disorders, or depressive disorders due to substances and/or medications, depressive disorders due to other medical problems, etc.);
* Patients with a cardiac pacemaker, cochlear implant, or other metal foreign body and any electronic equipment implanted in the body, patients with claustrophobia and other contraindications to magnetic resonance scanning, and patients with contraindications to rTMS treatment;
* History of epilepsy (presence of at least 2 uninduced seizures more than 24 hours apart, or diagnosis of the epileptic syndrome, or seizures within the past 12 months); Or currently received medications or other treatments that will lower the seizure threshold;
* History of ECT, rTMS, and light therapy within 3 months;
* Patients with serious heart, liver, kidney diseases, diabetes and other serious physical diseases, causing symptoms and signs of brain abnormalities, or body failure;
* Patients with organic brain diseases (such as ischemic stroke, cerebral hemorrhage, brain tumor, etc.) and a history of severe brain trauma as judged by the researcher;
* Female of childbearing potential who plans to become pregnant during the trial.
* Female that is pregnant or breastfeeding.
* Substance abuse or dependence (including alcohol, drugs, and other psychoactive substances) in the past 1 year;
* First-degree relatives have bipolar affective disorder.
* There is a significant risk of suicide (MADRS item 10 ≥ 5).
* Difficulty or inability to engage in normal communication, understand or follow instructions, and cooperate with treatment and evaluators.
* Currently participating in clinical trials of other drugs or physical therapy (e.g. deep brain stimulation (DBS), electroconvulsive therapy (ECT), rTMS).
* Investigators think that was inappropriate to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
change in MADRS | Baseline, Day 14(immediate post-treatment)
  A provider-administered questionnaire was used to assess remission and recovery from depression. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The MADRS has an overall score range from 0-60, with higher scores corresponding to higher levels of depression

SECONDARY OUTCOMES:
change in MADRS | Baseline, Day 7, Day 14, Day 21
  A provider-administered questionnaire was used to assess remission and recovery from depression. The MADRS is a ten-item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. The MADRS has an overall score range from 0-60, with higher scores corresponding to higher levels of depression
change in HAMD | Baseline, Day 7, Day 14, Day 21
  A provider-administered questionnaire was used to assess remission and recovery from depression. The Hamilton Depression Rating Scale (HAMD) is the most widely used clinician-administered depression assessment scale. The Ham-17 version consists of 17 items assessing mood, guilt, general somatic symptoms, work and activities, anxiety, and slowness of thought and speech. Each item is scored on a scale of 0 to 4, except for the somatic, sleep, and insight items which are scored 0 to 2. On the HAMD-17 there can be a total score of 52. Higher scores represent higher depression severity
cognitive change in Digit Symbol Substitution Test (DSST) | Baseline, Day 14(immediate post-treatment)
  Cognitive scores are measured using Chinese brief cognitive test (C-BCT), the DSST equires a subject to match symbols to numbers according to a key located on the top of the page
cognitive change in a continuous performance test (CPT） | Baseline, Day 14(immediate post-treatment)
  CPT from the C-BCT measures a person's sustained and selective attention
cognitive change in Trail-Making Test (TMT) | Baseline, Day 14(immediate post-treatment)
  The TMT test from the C-BCT can provide information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning
cognitive change in Digit Span Test (DST) | Baseline, Day 14(immediate post-treatment)
  DST from the C-BCT is a measure of verbal short term and working memory that can be used in two formats, Forward Digit Span and Reverse Digit Span

CONTACTS AND LOCATIONS:
Overall Officials: Hesheng Liu, Ph.D., Study Chair — Changping Laboratory
Locations (1):
- Henan Mental Hospital, Xinxiang, Henan, China